CLINICAL TRIAL: NCT06024408
Title: A Three-Part, Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ALN-PNP siRNA in Participants With Nonalcoholic Fatty Liver Disease (NAFLD) and a PNPLA3 Genetic Risk Factor
Brief Title: A Trial to Learn if Receiving ALN-PNP siRNA is Safe and Well Tolerated, and How it Works in Adult Participants With Nonalcoholic Fatty Liver Disease (NAFLD) and a Genetic Risk Factor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-PNP-NASH-2255
Record Dates: First submitted 2023-08-16; First posted 2023-09-06 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Nonalcoholic Fatty Liver Disease (NAFLD); Nonalcoholic Steatohepatitis (NASH); Genetic Risk Factor
Keywords: Homozygous; Heterozygous
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- Part A: Placebo (Placebo Comparator): Participants who are homozygous for the PNPLA3 rs738409:G risk allele will be randomized 1:1:1:1
  Interventions: Drug: Placebo
- Part A: Low Dose (Experimental): Participants who are homozygous for the PNPLA3 rs738409:G risk allele will be randomized 1:1:1:1
  Interventions: Drug: ALN-PNP
- Part A: Mid Dose (Experimental): Participants who are homozygous for the PNPLA3 rs738409:G risk allele will be randomized 1:1:1:1
  Interventions: Drug: ALN-PNP
- Part A: High Dose (Experimental): Participants who are homozygous for the PNPLA3 rs738409:G risk allele will be randomized 1:1:1:1
  Interventions: Drug: ALN-PNP
- Part B: Placebo (Placebo Comparator): Participants who are homozygous for the PNPLA3 rs738409:G risk allele will be randomized 1:1:1:1
  Interventions: Drug: Placebo
- Part B : Low Dose (Experimental): Participants who are homozygous for the PNPLA3 rs738409:G risk allele will be randomized 1:1:1:1
  Interventions: Drug: ALN-PNP
- Part B: Mid Dose (Experimental): Participants who are homozygous for the PNPLA3 rs738409:G risk allele will be randomized 1:1:1:1
  Interventions: Drug: ALN-PNP
- Part B: High Dose (Experimental): Participants who are homozygous for the PNPLA3 rs738409:G risk allele will be randomized 1:1:1:1
  Interventions: Drug: ALN-PNP
- Part C: Placebo (Optional) (Placebo Comparator): Sponsor may elect to enroll participants who are heterozygous for the PNPLA3 rs738409:G risk allele and may be randomized 1:1
  Interventions: Drug: Placebo
- Part C: High Dose (Optional) (Experimental): Sponsor may elect to enroll participants who are heterozygous for the PNPLA3 rs738409:G risk allele and may be randomized 1:1
  Interventions: Drug: ALN-PNP

INTERVENTIONS:
Drug: ALN-PNP — Part A: Administered as single subcutaneous (SC) injection on day 1 Part B and Part C: Administered SC every 12 weeks (Q12W x2)
  Arms: Part A: High Dose; Part A: Low Dose; Part A: Mid Dose; Part B : Low Dose; Part B: High Dose; Part B: Mid Dose; Part C: High Dose (Optional)
Drug: Placebo — Part A: Administered as single SC injection on day 1 Part B and Part C: Administered SC every 12 weeks (Q12W x2)
  Arms: Part A: Placebo; Part B: Placebo; Part C: Placebo (Optional)

SUMMARY:
This study is researching an experimental drug called ALN-PNP. This study is focused on participants who are known to have nonalcoholic fatty liver disease (NAFLD), and a specific variant of the patatin-like phospholipase domain containing 3 (PNPLA3) gene.

The aim of this study is to see how safe, tolerable, and effective the study drug is.

This study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How the study drug works to change liver fat content in NAFLD
* How much study drug and study drug metabolites (byproduct of the body breaking down the study drug) are in your blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)
* Better understanding of the study drug and NAFLD

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants from 18 (or country's legal age of adulthood) to 65 years of age, inclusive, at screening visit 1
2. Body mass index (BMI) from 23.0 kg/m^2 to 40.0 kg/m^2, inclusive, for East Asians (including but not limited to South Koreans, Chinese, Taiwanese, and Japanese) and BMI from 27.0 kg/m^2 to 40.0 kg/m^2, inclusive, for any other ethnicity at screening visit 1
3. Meets genotype criteria for the rs738409:G PNPLA3 risk allele: homozygotes (for Part A and Part B) or heterozygotes (optional Part C); p.I148M variant (PNPLA3 rs738409:G [p.I148M]) at screening visit 1
4. Liver fat content ≥8.5% as measured by MRI-PDFF at screening visit 3
5. Generally stable diet (based on participant's recall) for at least 3 months prior to the screening visit

Key Exclusion Criteria:

1. Evidence of other forms of known chronic liver disease, as defined in the protocol
2. Has a contraindication to MRI examinations, such as persons with cardiac pacemaker and implants made out of metal (for example, cochlear implant, nerve stimulators, magnetic vascular clips, and metallic heart valve), severe claustrophobia, or other contraindications for MRI
3. Is taking a medication to treat a co-morbid condition that is not permitted during the study
4. Has any laboratory parameter assessments at screening, as defined in the protocol
5. History of Type 1 diabetes
6. Bariatric surgery within approximately 5 years prior or planned during the study period
7. Has lost or gained more than 4.0% body weight over the 3 months prior to or during the screening period
8. Has known human immunodeficiency virus (HIV) infection, evidence of current or chronic hepatitis B virus (HBV) infection, or current or chronic hepatitis C virus (HCV) infection, as defined in the protocol
9. Was hospitalized (ie, >24 hours) for any reason within 30 days of the screening visit

Note: Other protocol defined Inclusion/Exclusion Criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 253 days
Severity of TEAEs | Up to 253 days

SECONDARY OUTCOMES:
Change in liver fat fraction by magnetic resonance imaging proton density fat fraction (MRI-PDFF) in participants with NAFLD | Baseline up to 253 days
Change in low-density lipoprotein cholesterol (LDL-C) in participants with NAFLD | Baseline up to 253 days
Change in high-density lipoprotein cholesterol (HDL-C) in participants with NAFLD | Baseline up to 253 days
Change in triglycerides (TG) in participants with NAFLD | Baseline up to 253 days
Change in lipoprotein a (Lp(a)) in participants with NAFLD | Baseline up to 253 days
Change in apolipoprotein A1 (ApoA1) in participants with NAFLD | Baseline up to 253 days
Change in apolipoprotein B (ApoB) in participants with NAFLD | Baseline up to 253 days
Concentration of ALN-PNP and potential major metabolite(s) in plasma over time | Up to 253 days
Incidence of anti-drug antibodies (ADAs) to ALN-PNP | Up to 253 days
Titer of anti-drug antibodies (ADAs) to ALN-PNP | Up to 253 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (5):
- South Korea (5):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheong Buk-do
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/